CLINICAL TRIAL: NCT03293849
Title: A Patient Navigation Program to Increase Access to Early Supportive Care in Patients With Stage IV Solid Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Global Cancer Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REF. 2191
Record Dates: First submitted 2017-09-06; First posted 2017-09-26 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2019-07

CONDITIONS: Neoplasm Metastasis
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Navigation Arm (Experimental): After an assessment of supportive care needs, a patient navigator will present assessment results and develop and implement a personalized supportive care intervention plan based on the findings in collaboration with a multidisciplinary supportive care team, formed by oncologists and pain and palliative care specialists. The developed plan will be sent to the treating oncologist and oncology team.
  Interventions: Other: Patient Navigation
- Control Arm (No Intervention): Assessment results will be provided in printed and electronic form to the treating oncologist for their review. Referrals or interventions for patients allocated to the control arm will be coordinated by the treating oncologist without involvement from the patient navigator or the study team.

INTERVENTIONS:
Other: Patient Navigation — The patient navigator will discuss the results and supportive care recommended interventions of the multidisciplinary team with the patient. Those interventions which are accepted by patient are initiated when possible, and referrals are made as planned. The study patient navigator will review advance directive planning with those patients who are candidates to complete an advanced directive under Mexican law, and will facilitate the resources to complete the advance directive.
  Arms: Patient Navigation Arm

SUMMARY:
In this randomized clinical trial, patients with Stage IV solid tumors will be enrolled in a patient navigator-led generalist palliative and supportive care intervention or in usual care led by their treating physician. The patient navigator will assess the patient's palliative and supportive care needs using standardized quality of life and symptoms questionnaires and present this assessment to a multidisciplinary team composed of oncologists and palliative care specialist. The multidisciplinary team will develop a personalized supportive care plan for the patient which will then be presented and discussed by the patient navigator. Those interventions which are accepted by the patient will be implemented by the patient navigator, who will also provide education and teaching. The patient navigator will also help eligible patients complete advanced directives according to local rules and regulations. The patient navigator will follow the patients both in person and by telephone to ensure that the recommended interventions have been implemented. Three months after enrollment the patients will undergo quality of life and symptom assessment once again, and the implementation of interventions will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years of age and older
2. Newly diagnosed stage IV solid tumor
3. Recurrent stage IV solid tumor

Exclusion Criteria:

1. Homeless persons
2. History of drug abuse or alcoholism
3. Patients suffering from major psychotic disorders or uncontrolled psychiatric disorders
4. Mentally disabled patients
5. Incarcerated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Referrals to Supportive Care Services | Three months
  Proportion of patients who agree to participate in the patient navigation program, complete the initial assessment, meet with the patient navigator to discuss advanced care planning and supportive care interventions and obtain the appropriate referrals and consultations.

SECONDARY OUTCOMES:
Rate of advanced directive completion | Three months
  Obtaining a signed advanced directive
Implementation of planned supportive care interventions | Three months
  Documentation of the planned interventions on the patient's medical record at end-of-study
Changes in QOL | Three months
  Changes in QOL measured using the FACT-G from baseline.
Changes in self-reported pain | Three months
  Changes in self reported pain measured using the BPI scale from baseline.
Use of chemotherapy at the end of life | 18 months
  Interval between last administration of chemotherapy and death
Healthcare utilization | 18 months
  Sum of hospital admissions, emergency room admissions and ICU admissions during the study period
Survival | 18 months
  Overall survival (defined as time from study enrollment to last recorded visit or death)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Soto Perez de Celis, MD, MSc, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided